CLINICAL TRIAL: NCT04416438
Title: Observational Study of the Impact of the COronaVirus Disease 2019 (COVID-19) Epidemic on Patients With Myeloproliferative Neoplasias
Brief Title: COVID-19 Epidemic and Patients With Myeloproliferative Neoplasias
Acronym: COVIM
Status: Completed | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: French Intergroup of Myeloproliferative syndromes (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVIM
Record Dates: First submitted 2020-06-03; First posted 2020-06-04 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Myeloproliferative Neoplasm; COVID-19 Infection
MeSH Terms: conditions — Myeloproliferative Disorders; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The classic myeloproliferative neoplasias (MNP), including polycythemia vera (PV), essential thrombocythemia (ET), primary myelofibrosis (PMF) or secondary to PV or ET, are among the most frequent of malignant hemopathies, with overall prevalence estimated at around 10,000 patients followed in France. Due to the median age of patients around 65, the frequency of cardiovascular complications of these thrombogenic diseases and the impact of cytoreductive treatments on immune cells, these patients are considered to be at risk of developing forms severe of COVID-19. This study will assess the impact of MNPs on the risk of developing a severe form of COVID-19, identify new risk factors linked to the disease as well as the impact of treatments for MNPs according to their pharmacological class.

DETAILED DESCRIPTION:
It is a descriptive, prospective epidemiological study using retrospective patient data, multicenter, non-interventional, carried out in FIM (French Intergroup of Myeloproliferative syndromes) / FILO (French Innovative Leukemia Organization) centers.

This is an exploratory descriptive study in order to put in place as soon as possible a possible strategy for the protection of patients most at risk.

The study will include all consecutive patients with MNP according to the WHO (World Health Organization) classification seen in consultation or teleconsultation over the duration of the study, whether or not they have had a COVID-19 infection.

The collection of clinical data, treatment regimens and survival and death data will be carried out by the investigator or a member of his medical team, after delivering an information note to the patient informing him of the computerized processing of his data, subject to the patient's non-objection.

The diagnosis of asymptomatic COVID 19 will be made on the presence of a positive serology and on the absence of clinical signs on questioning.

The presence of a symptomatic COVID 19 infection will be posed on the presence of clinical signs +/- CT as identified by the practitioner who treated the patient and confirmed or not by a positive PCR and / or a positive serology.

Data collected:

* Socio-demographic data (gender, date of birth)
* Description of hemopathy and its treatment
* Description of COVID-19 infection and its management
* Biological data: blood count, specific COVID-19 test results if available (PCR, serology).
* History, comorbidities
* Evolution of COVID-19 infection and possible specific treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient with PV, ET, PMF or MF secondary to PV or ET diagnosed before the COVID-19 pandemic
* Seen in consultation or teleconsultation from May 2020 or deceased if the investigator became aware of this death during the study period

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Classic myeloproliferative neoplasias (MPN), including polycythemia vera (PV), essential thrombocythemia (ET), primary myelofibrosis (PMF) or secondary to PV or ET, and infected by COVID-19
Sampling Method: Probability Sample
Enrollment: 1793 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of serious coronavirus infection in different MNP patient subgroups | Through inclusion period, an average of 6 months
  The crude rate of cumulative incidence of serious infection proven to COVID-19, compared to the population of the same age, same sex, same region of residence during the epidemic period.
Proportion of MNP patients who had COVID-19 infection during the 2020 epidemic. | Through inclusion period, an average of 6 months
  Number of MNP patients who had COVID-19 compared to general population in France
Rate of death of MNP patients who had COVID-19 | Through study completion, an average of 1 year
  Number of MNP patients who died from COVID-19
Rate of passages in intensive care with need for mechanical ventilation | Through study completion, an average of 1 year
  Number of MNP patients hospitalized in intensive care with need for mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques KILADJIAN, Pr, Principal Investigator — FIM; Laurence LEGROS, Dr, Principal Investigator — FIM
Locations (1):
- Paris Saint Louis, Paris, France